CLINICAL TRIAL: NCT00866593
Title: A Randomized Double-blind Parallel Innovator-Controlled Multicenter Clinical Trial to Evaluate the Efficacy and Safety of Generic Escitalopram Oxalate Tablets in the Treatment of Chinese Patients With Depression
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of Generic Escitalopram in Depression
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Jiangsu Nhwa Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004L04118; SMHC-101
Record Dates: First submitted 2009-03-18; First posted 2009-03-20 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Depression
Keywords: major depressive disorder(MDD); depression; antidepressant; escitalpram oxalate; generic; innovator; Lexapro; efficacy; safety; multicenter; double-blind; randomized; chinese; HAMD; MADRS; HAMA; VAS-PI; SDS; CGI
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Generic Escitalopram Oxalate Tablets
  Interventions: Drug: Generic Escitalopram
- 2 (Active Comparator): Innovator Escitalopram(Lexapro®)
  Interventions: Drug: Innovator Escitalopram

INTERVENTIONS:
Drug: Generic Escitalopram — 10mg/d or 20mg/d
  Other Names: Generic Escitalopram Oxalate Tablet
  Arms: 1
Drug: Innovator Escitalopram — 10mg/d or 20mg/d
  Other Names: Lexapro®
  Arms: 2

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of Generic Escitalopram in the treatment of Chinese patients with depression compared with Innovator Escitalopram(Lexapro®) by evaluating the change of HAMD-17 total score from the baseline to week 8.

DETAILED DESCRIPTION:
This is a double-blind, parallel assignment, randomized and innovator controlled study. The subjects investigated are outpatients with major depressive disorder(MDD)according to DSM-IV from the Chinese population. The screening phase lasts for 1 week. The eligible patients enter the next randomized treatment phase. The fixed dose(generic escitalopram 10mg/d or Innovator Escitalopram(Lexapro®) 10mg/d) duration is 2 week. After the first 2 weeks, according to CGI and investigator's assessment the patients are administrated 2 different dose, one is previous dose 10mg/d, the other is high dose 20mg/d. In this study, total duration lasts for 8 weeks.

The efficacy and safety of Innovator Escitalopram(Lexapro®) in the treatment of patients with MDD have been confirmed by multiple double blind studies. This study is designed to evaluate the efficacy and safety of genetic escitalopram in the treatment of Chinese patients with MDD. Therefore, the double blind and innovator control(Lexapro®) design should be selected for this study. The drug titration method and dose are within the range specified in the instruction and patients with MDD are tolerant to the drug in practical clinical treatment.

The purpose of MDD patient treatment is to improve the core symptoms, prevent suicide, alleviate the side reactions caused by the antidepressant, and recover the life functions of patients. Generally, the treatment in the acute phase lasts for 6 to 8 weeks. In this study, the treatment in the acute phase lasts for 8 weeks.

The rating scales used in this study are standard psychiatric rating scales with good validity and are widely used in the study of antidepressants and in the treatment of patients with MDD. The high inter-investigator reliability and repeated measurement reliability of these scales(HAMD,MADRS,HAMA) have been proved by multiple studies. The clinical global impression (CGI) is a simple but convenient global impression scale. It is applicable to any patients treated and studied by the psychiatric department. The VAS-PI(Visual Analog Scale-Pain Intensity) is used to evaluate the reduction in pain intensity,a common symptom of patients with MDD. It has good reliability and validity. The Sheehan Disability Scale (SDS) was developed to assess functional impairment in three inter-related domains; work/school, social and family life.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* Patients who met DSM-IV criteria for major depressive disorder(MDD):a single major depressive episode or recurrent major depressive episode, without psychotic features, MDD is primary mental disorder
* Age from 18-65 years old, male or female
* HAMD-17 total score at least 20 at screening and baseline, and first item's score at least 2
* CGI-S at least 4 at screening and baseline
* Written informed consent provided by patient himself/herself

Exclusion Criteria:

* Severe suicide attempt
* Any unstable medical illness would affect study or increase patients' risk to participate this study, including disease of heart, lung, liver, kidney,cardiovascular system, eyes, nervous system, endocrine system, hematological system etc.
* History of epilepsy(except children febrile seizure/convulsion)
* Known history of high intraocular pressure or angle closure glaucoma
* Psychoactive substance abuse or dependence within 1 year prior enrollment
* Depressive episode due to other mental disorders or physical diseases
* Bipolar disorder, rapid cycling/circulation
* Female patients during their pregnant and lactation period or childbearing potential during study
* History of severe drug hypersensitivity
* A significantly clinical abnormal value in ECG or lab results which would affect assessment for efficacy or safety decided by the investigator
* ALT and AST values in the liver function test exceeding two times of the upper limits of normal values
* Participation in another drug trial within 28 days prior enrollment into this study
* Use of MAOI within 4 weeks prior to randomization
* Duration of discontinuing other psychotropics is shorter than its 7 half life periods
* Patients can not administrate drug according to medical order
* HAMD total score decreased more than 25% from screening to baseline
* Use of Electroconvulsive therapy within half year prior enrollment
* Known lack of efficacy to escitalpram by formal treatment before
* Other situation unsuitable to enroll in this study as judged by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
the change of HAMD-17 total score | from the baseline to week 8

SECONDARY OUTCOMES:
the change of MADRS total score | from the baseline to week 8
the change of HAMA total score | from the baseline to week 8
the clinical global impression (CGI),including CGI-I and CGI-S | from the baseline to week 8
the change of VAS-PI | from the baseline to Week 8
the change of Sheehan Disability Scale(SDS) | from the baseline to Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Huafang LI, MD,PhD, Principal Investigator — Drug Clinical Trial Office, Shanghai Mental Health Center
Locations (6):
- China (6):
  - Hebei Mental Health Center, Baoding, Hebei
  - Nanjing Brain Hospital, Nanjing, Jiangsu
  - the First Affiliated Hospital，Medical School of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Xi'an Mental Health Center, Xi'an, Shaanxi
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - The First Affilliated Hospital Of Kunming Medical College, Kunming, Yunnan

REFERENCES:
- [Derived] Yu Y, Li H, Wang B, Li K, Xu X, Shi J, Gao C, Tan Q. Efficacy and safety of generic escitalopram versus Lexapro in the treatment of major depression: a multicenter double-blinded randomized controlled trial. Shanghai Arch Psychiatry. 2013 Apr;25(2):107-15. doi: 10.3969/j.issn.1002-0829.2013.02.007. PMID 24991142